CLINICAL TRIAL: NCT02857647
Title: The Effects of an Information Video on Anxiety and Bariatric Surgery Knowledge Among Bariatric Surgery Candidates
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assuta Medical Center (Other)
Responsible Party: Principal Investigator, Shiri Sherf Dagan, Shiri Sherf Dagan, Assuta Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0041-16
Record Dates: First submitted 2016-08-03; First posted 2016-08-05 (Estimated); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Bariatric Surgery Candidates
Keywords: Bariatric surgery; Anxiety; Nutrition knowledge; Weight loss expectations
MeSH Terms: conditions — Anxiety Disorders

ARMS (2):
- The experimental group (Experimental): Participants who will assigned to the experimental group will be asked to watch an information video of 30 minutes 1-2 weeks prior to the surgery date.
  n=100.
  Interventions: Behavioral: An information video
- The control group (No Intervention): Participants who will assigned to the control group will receive standard care and will not asked to watch a videotaped lecture prior to the surgery.
  n=100.

INTERVENTIONS:
Behavioral: An information video — Participants who will assigned to the experimental group will be asked to watch a 30 minutes videotaped lecture 1-2 weeks prior to the surgery date. Topics includes: types of surgeries, preparation to the hospitalization process and to the surgery (e.g. what to expect, personal equipment needs, description of the surgery admission process, etc.), dietary guidelines pre- and post-surgery (e.g. low carb diet 2-3 week prior to the surgery, post-surgery diet progression, techniques of eating and drinking, recommended dietary supplements), recommendation and tips for long term surgery success (e.g. definition of weight loss expectations, physiological, nutritional and life-style strategies for long-term weight loss).
  Arms: The experimental group

SUMMARY:
An interventional prospective study on 200 bariatric surgery candidates from the Assuta Medical Center (AMC). The first 100 patients will be assigned to the control group and the later 100 patients will be assigned to the experimental group. All the participants will receive standard care, and only those participants who will assigned to the experimental group will be asked to watch a videotaped lecture of 30 minutes 1-2 weeks prior to the surgery date. The videotaped lecture will include information and guidelines of bariatric surgery preparation. All participants will complete Bariatric surgery knowledge questionnaire and The state-trait anxiety inventory (STAI) questionnaire at the bariatric committee and once again at the pre-surgery clinic which take place 1-10 days pre-surgery.In addition, 20 participants will be recruited to a pilot study for the validation of the Bariatric surgery knowledge questionnaire.

DETAILED DESCRIPTION:
Only few studies have investigated anxiety level, bariatric surgery and nutrition knowledge and weight loss expectations prior to bariatric surgery. No studies have been published on how preparation lectures prior to bariatric surgery impact on anxiety level and on patients' knowledge. A better preparation process prior to the bariatric surgery may have an impact on higher success rates of bariatric surgeries.

Our study is an interventional prospective study on 200 bariatric surgery candidates from the Assuta Medical Center (AMC). The first 100 patients will be assigned to the control group and the later 100 patients will be assigned to the experimental group. All the participants will receive standard care, and only those participants who will assigned to the experimental group will be asked to watch a videotaped lecture of 30 minutes 1-2 weeks prior to the surgery date. The videotaped lecture will include information and guidelines of bariatric surgery preparation. Topics includes: types of surgeries, preparation to the hospitalization process and to the surgery (e.g. what to expect, personal equipment needs, description of the surgery admission process, etc.), dietary guidelines pre- and post-surgery (e.g. low carb diet 2-3 week prior to the surgery, post-surgery diet progression, techniques of eating and drinking, recommended dietary supplements), recommendation and tips for long term surgery success (e.g. definition of weight loss expectations, physiological, nutritional and life-style strategies for long-term weight loss). All participants will complete Bariatric surgery knowledge questionnaire and The state-trait anxiety inventory (STAI) questionnaire at the bariatric committee and once again at the pre-surgery clinic which take place 1-10 days pre-surgery. In addition, 20 participants be recruited to a pilot study for the validation of the Bariatric surgery knowledge questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Pre-surgery: 18 years old or older, BMI > 40 kg/m² or BMI > 35 kg/m² with comorbidities and approval of the AMC committee to undergo bariatric surgery.
* Surgery types: laparoscopic sleeve gastrectomy (LSG), Roux-en-Y gastric bypass (RYGB) and Single-anastomosis gastric bypass (SAGB)
* Surgery will take place at Assuta medical center.
* Reading and speaking Hebrew.

Exclusion Criteria:

* Previous bariatric surgery.
* Surgery types: laparoscopic adjustable gastric band (LAGB) or biliopancreatic diversion with duodenal switch (BPD-DS)
* Less than 2 weeks between bariatric committee and surgery date

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Anxiety | pre-surgery
  Pre-surgery anxiety level will be measured by the state-trait anxiety inventory (STAI) questionnaire.

SECONDARY OUTCOMES:
Bariatric surgery and nutrition knowledge | pre-surgery
  Bariatric surgery and nutrition knowledge will be measured by a questionnaire written by investigators.
Weight loss expectation | pre-surgery

REFERENCES:
- [Derived] Sherf-Dagan S, Hod K, Mardy-Tilbor L, Gliksman S, Ben-Porat T, Sakran N, Zelber-Sagi S, Goitein D, Raziel A. The Effect of Pre-Surgery Information Online Lecture on Nutrition Knowledge and Anxiety Among Bariatric Surgery Candidates. Obes Surg. 2018 Jul;28(7):1876-1885. doi: 10.1007/s11695-018-3134-y. PMID 29455404